CLINICAL TRIAL: NCT00471419
Title: Phase II Study of AL-2178 (FID 109980) in the Treatment of Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-31
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2008-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — rimexolone

INTERVENTIONS:
Drug: Rimexolone

SUMMARY:
The purpose of this study is to see if Rimexolone (FID 109980) is a safe and effective treatment of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* documented dry eye history
* ocular symptoms
* tear use
* dry eye ocular signs

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Corneal staining; dry eye sympton | Immediate

SECONDARY OUTCOMES:
Corneal staining; dry eye sympton | Prolonged

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brubaker, PhD, Study Director — Alcon Research
Locations (1):
- Cleveland, Cleveland, Ohio, United States